CLINICAL TRIAL: NCT01578681
Title: Multicenter Randomized Placebo-controlled Trial to Evaluate the Efficacy of the ELTGOL Technique in the Drainage of Secretions in Patients With Bronchiectasis
Brief Title: ELTGOL and Bronchiectasis. Respiratory Therapy
Acronym: ELTGOLBQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Dr. Montserrat Vendrell Relat, Pneumology Doctor, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08/10
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Respiratory; Complications, Therapy; Bronchiectasis
Keywords: bronchiectasis; respiratory therapy; airway clearance
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Airway clearance, bronchiectasis (Active Comparator): The patient would be selected randomly to one of the two groups (intervention or placebo). And follow up for one year with regular visits with the physician and the respiratory therapist.
  Each patient will be visited 7 times. At each visit all the variable will be registered. Patient will have also a personal registration diary.
  Interventions: Procedure: Low Expiration Open glottis inferolateral (ELTGOL)
- bronchiectasis, stretching (Placebo Comparator): The patient would be selected randomly to one of the two groups (intervention or placebo). And follow up for one year with regular visits with the physician and the respiratory therapist.
  Each patient will be visited 7 times. At each visit all the variable will be registered. Patient will have also a personal registration diary.
  Interventions: Procedure: Stretching

INTERVENTIONS:
Procedure: Low Expiration Open glottis inferolateral (ELTGOL) — Place the affected lung in infralateral, asks the patient to make an inspiration without being forced to medium volume, and then a slow expiration with the glottis open, down to residual volume. If the therapist is present place the abdominal caudal hand at putting pressure cranial head and hand is placed over the rib cage at a pressure of closing the rib cage. Otherwise, the patient self-administered intertwining arms and abdominal rib at top exerting the same pressure. In case you have two lungs affected the art will take place on one side and then the opposite.
  Other Names: airway clearance
  Arms: Airway clearance, bronchiectasis
Procedure: Stretching — Patient will be instructed to do muscle stretching of the thorax
  Arms: bronchiectasis, stretching

SUMMARY:
The ELTGOL technique improves mucociliary clearance in adult patients with bronchiectasis.

Primary objective:

-To evaluate the efficacy of ELTGOL in stable state patients with bronchiectasis compared to placebo.

Secondary objectives:

* To evaluate the level of knowledge of airway clearance techniques and adherence to them in patients with bronchiectasis.
* To assess the side effects during the procedure: oxygen desaturation, increased dyspnea and hemoptysis.

DETAILED DESCRIPTION:
The incidence of bronchiectasis has increased in recent years resulting in greater costs, including periods of hospitalisation and the prescription of drugs.

The mucociliary clearance mechanism is impaired in these patients, and chest physiotherapy has been recommended for patients with bronchiectasis and chronic productive cough and/or evidence of mucus plugging on HRCT.

However, to date, there is insufficient evidence of benefits of chest physiotherapy through randomised controlled trials. Furthermore it rests unclear the most effective technique, the frequency and optimum duration of the RP and the most suitable variables to monitor.

A multicenter clinical trial into the efficacy of one chest physiotherapy technique in airway clearance will fill this important "gap" in the scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

* All subjects ≥ 18 years old.
* Diagnosis of bronchiectasis using a high-resolution computed tomography (HRCT) chest scan performed in the last 2 years.
* Clinically stable disease (defined as no requirement for antibiotics for exacerbation in the 4 weeks preceding study entry.
* Chronic sputum expectoration >10ml/24h.

Exclusion Criteria:

* Bronchiectasis secondary to cystic fibrosis.
* Inability to perform physiotherapy techniques.
* Inability to attend the following controls.
* Treatment with mucolytics, DNase or hypertonic saline during the study.
* Smokers and ex-smokers ≥ 10 pack/year.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of ELTGOL in stable state patients with bronchiectasis compared to placebo | 1 year
  The primary endpoint for the study is:
  •Sputum volume during the procedure in the second visit and 24h post treatment which is defined as the volume of mucus expectorated during the physiotherapy procedure and 24h post treatment measured by ml.

SECONDARY OUTCOMES:
Side effects, knowledge | 1 year
  * To evaluate the level of knowledge of airway clearance techniques and adherence to them in patients with bronchiectasis.
  * To assess the side effects during the procedure: oxygen desaturation, increased dyspnea and hemoptysis.

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat V Relat, Doctor, Principal Investigator — Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Locations (1):
- Hospital Universitari Dr. Josep Trueta, Girona, Spain

REFERENCES:
- [Derived] Munoz G, de Gracia J, Buxo M, Alvarez A, Vendrell M. Long-term benefits of airway clearance in bronchiectasis: a randomised placebo-controlled trial. Eur Respir J. 2018 Jan 11;51(1):1701926. doi: 10.1183/13993003.01926-2017. Print 2018 Jan. PMID 29326318